CLINICAL TRIAL: NCT04940377
Title: Postoperative Venous Thromboembolism Risk in 140,831 Surgical Patients - a Genetic Association Cohort Study
Brief Title: Effect of the Genotype on Postoperative DVT
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Martin Sillesen, Assoc. Prof., Rigshospitalet, Denmark
Other Study IDs: 60861
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative Venous Thromboembolism Events (VTE) constitute a major source of morbidity and mortality after surgery. The aim of this study was to investigate whether commonly occurring Single Nucleotide Polymorphisms (SNPs) are associated with VTE in the surgical setting.

DETAILED DESCRIPTION:
Data extracted from the participants in the UK Biobank collaborative study. Two cohorts will be examined:

1. Surgical cohort, consisting of all patients with a registered surgical procedure in the UK biobank repository
2. Validation cohort, consisting of all non-surgical patients in the UK biobank repository.

A GWAS approach will be used to associated commonly occurring single nucleotide polymorphisms (SNPs) with a postoperative venous thromboembolic event (VTE) within 30 days of a surgical procedure in the surgical cohort.

Findings from the surgical GWAS step will be replicated in the Validation cohort in order to assess whether the same SNPs drive both surgical and non-surgical VTE risk.

A final GWAS model will be fielded, correction for confounders including sex, age, smoking, obesity and open/minimal invasive surgery (surgical discovery GWAS only).

ELIGIBILITY:
Inclusion Criteria:

- All patients included in the UK biobank repository

Exclusion criteria:

- None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers followed by the UK biobank consortium
Sampling Method: Non-Probability Sample
Enrollment: 502505 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Postoperative VTE event | 30 days of a surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark